CLINICAL TRIAL: NCT02176902
Title: A Phase II Randomized, Open-Label, Two-Arm Study of a Low Omega-6, High Omega-3 Fat Diet Combined With Fish Oil vs. a Control Group in Men on Active Surveillance for Prostate Cancer
Brief Title: Low-Fat Diet and Fish Oil in Men on Active Surveillance for Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pharmavite LLC (Industry); Seafood Industry Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-000432; NCI-2014-01257 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-000432 (Other: Jonsson Comprehensive Cancer Center); P50CA092131 (NIH)
Record Dates: First submitted 2014-06-23; First posted 2014-06-27 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2024-08

CONDITIONS: Adenocarcinoma of the Prostate; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (control) (No Intervention): Patients receive no intervention.
- Arm II (fish oil) (Experimental): Patients receive dietary counseling with research dietitian weekly for 1 month and then monthly for 11 months. Patients are given guidelines with recommended meals to follow a low omega-6, high omega-3 fat diet combined with fish oil. Patients also receive 4 fish oil capsules per day PO for 1 year.
  Interventions: Behavioral: behavioral dietary intervention; Dietary Supplement: omega-3 fatty acid; Other: laboratory biomarker analysis

INTERVENTIONS:
Behavioral: behavioral dietary intervention — Receive dietary counseling
  Arms: Arm II (fish oil)
Behavioral: behavioral dietary intervention — Receive guidelines for low-fat diet
  Arms: Arm II (fish oil)
Dietary Supplement: omega-3 fatty acid — Given PO
  Other Names: fish oil; n-3 fatty acid; O3FA
  Arms: Arm II (fish oil)
Other: laboratory biomarker analysis — Correlative studies
  Arms: Arm II (fish oil)

SUMMARY:
This randomized phase II trial will evaluate if a low omega-6, high omega-3 fat diet combined with fish oil has the potential to delay disease progression in patients with prostate cancer undergoing active surveillance.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if a 1-year low omega-6, high omega-3 fat diet combined with fish oil results in decreased prostate cancer Ki-67 index as compared to a control group in men on active surveillance.

SECONDARY OBJECTIVES:

I. Evaluate the effect of a low-fat (LF)/fish oil (FO) intervention on prostate biopsy tissue markers of progression, prostate biopsy pathologic features (Gleason grade, tumor volume ), prostate-specific antigen (PSA), and long-term clinical outcomes (clinical progression, prostate cancer therapies).

II. Evaluate potential surrogate biomarkers of proliferation (red blood cell [RBC] membrane fatty acid analyses, ex-vivo bioassay).

III. Determine if a correlation exists between free fatty acid receptor 4 (GPR120) levels and progression markers in response to the LF/FO intervention.

IV. Evaluate effect of the intervention on the National Comprehension Cancer Network (NCCN) risk group V. Evaluate compliance with a 1-year + 2 year extension LF/FO intervention. VI. Evaluate safety of a 1-year + 2-year extension LF/FO intervention.

OUTLINE: Patients are randomized to 1 of 2 arms. ARM I: Patients receive no intervention.

ARM II: Patients receive dietary counseling with a research dietitian weekly for 1 month and then monthly for 11 months. Patients are given guidelines with recommended meals to follow a high omega-3, low omega-6 diet comprising 30% kilocalories (Kcal) from fat, 15% Kcal from protein, and 65% Kcal from carbohydrates for 1 year. Patients also receive 4 fish oil capsules per day orally (PO) for 1 year.

After completion of study, patients are followed up yearly for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients sign the informed consent
* Patient had a prostate biopsy performed by Dr. Mark with the Artemis device and has adenocarcinoma of the prostate
* Patient elects to undergo active surveillance
* Clinical stage T2c or less
* Gleason grade 3+4 or less
* PSA < 25
* Geographically able to have study visits at the University of California, Los Angeles (UCLA) Clinical Research Unit
* Subjects are willing to not consume lycopene, green tea or pomegranate supplements or pomegranate juice during the 1-year study
* If subjects are randomized to the control group they agree to not consume fish oil capsules during the 1-year study

Exclusion Criteria:

* Diagnostic prostate biopsy with only 1 core with cancer and < 5% of tissue from that core involved with cancer
* Patient has taken finasteride or dutasteride during the prior year
* Patient has taken fish oil during the prior 3 months
* Patient had prior treatment for prostate cancer (surgery, radiation, local ablative therapy, anti-androgen therapy or androgen deprivation therapy)
* Patient has other medical conditions that exclude him from undergoing a repeat prostate biopsy at 1-year
* Patient has allergy to fish

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Ki-67 index | 1 year
  The primary statistical analysis will be to compare the Ki67 index between the two intervention arms using a negative binomial mixed effects model

SECONDARY OUTCOMES:
Composite measure: Prostate biopsy tissue markers of proliferation, cell cycle progression, and prostate biopsy pathologic features (Gleason grade, percent of cores with cancer, and percent of tissue with cancer) | 1 year
  Different types of regression models will be used to assess the influence of the intervention and clinical characteristics (ex. logistic regression, ordinal regression, Poisson regression instead of linear regression).
Serum PSA | Up to 1 year
  Different types of regression models will be used to assess the influence of the intervention and clinical characteristics (ex. logistic regression, ordinal regression, Poisson regression instead of linear regression).
Composite measure: Long-term clinical outcomes (clinical progression, prostate cancer therapies) | Up to 15 years
  Different types of regression models will be used to assess the influence of the intervention and clinical characteristics (ex. logistic regression, ordinal regression, Poisson regression instead of linear regression).
Composite measure: Potential surrogate biomarkers of proliferation (RBC membrane fatty acid analyses, ex-vivo bioassay) | Up to 1 year
  Different types of regression models will be used to assess the influence of the intervention and clinical characteristics (ex. logistic regression, ordinal regression, Poisson regression instead of linear regression). Whether the omega-6/omega-3 ratio provides additional predictive information beyond group will be assessed by investigating whether it correlates with Ki-67 within each group.
Correlation of GPR120 expression in peripheral blood mononuclear cells (PBMCs) and prostate biopsy tissue with immunostaining of Ki67 and Decipher Score | Up to 1 year
  Linear regression will be used to correlate PBMC and biopsy GPR120 gene and protein expression to 1-year Ki-67 index and Decipher score . GPR120 gene and protein expression will be added to the linear regression for Ki-67 constructed with group and clinical/demographic covariates.
Compliance, defined as having taken 80% or more of the daily fish oil throughout the trial determined based on pill count | Up to 1 year
  Analysis of subject compliance to dietary regimen
Incidence of adverse events graded according to National Cancer Institute Common Toxicity Criteria version 4.0 | Up to 1 year
  Measure of adverse events incidence
Sample storage for future research | Up to 1 year
  Urine, plasma and flash frozen prostate tissue will be stored for future research evaluating the effects of a LF/FO diet on prostate cancer progression.

CONTACTS AND LOCATIONS:
Overall Officials: William Aronson, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Aronson WJ, Grogan T, Liang P, Jardack P, Liddell AR, Perez C, Elashoff D, Said J, Cohen P, Marks LS, Henning SM. High Omega-3, Low Omega-6 Diet With Fish Oil for Men With Prostate Cancer on Active Surveillance: The CAPFISH-3 Randomized Clinical Trial. J Clin Oncol. 2025 Mar;43(7):800-809. doi: 10.1200/JCO.24.00608. Epub 2024 Dec 13. PMID 39671538